CLINICAL TRIAL: NCT06138470
Title: Evaluation of the Effect of a Combination of Plants (saffron and Scutellaria) to Regulate Mood
Brief Title: Evaluation of the Effect of a Combination of Plants to Regulate Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comercial Quimica Masso, S.A (Industry)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SAFFRUP
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Mood Regulation
MeSH Terms: interventions — Scutellaria baicalensis extract; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Saffron extract (Active Comparator)
  Interventions: Dietary Supplement: Saffron extract
- Scutellaria baicalensis extract (Active Comparator)
  Interventions: Dietary Supplement: Scutellaria baicalensis extract
- Saffron and Scutellaria baicalensis extract (Active Comparator)
  Interventions: Dietary Supplement: Saffron and Scutellaria baicalensis extract
- Placebo (maltodextrin) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (maltodextrin)

INTERVENTIONS:
Dietary Supplement: Saffron extract — Food supplements are taken during 6 weeks by healthy volunteers
  Arms: Saffron extract
Dietary Supplement: Scutellaria baicalensis extract — Food supplements are taken during 6 weeks by healthy volunteers
  Arms: Scutellaria baicalensis extract
Dietary Supplement: Saffron and Scutellaria baicalensis extract — Food supplements are taken during 6 weeks by healthy volunteers
  Arms: Saffron and Scutellaria baicalensis extract
Dietary Supplement: Placebo (maltodextrin) — Food supplements are taken during 6 weeks by healthy volunteers
  Arms: Placebo (maltodextrin)

SUMMARY:
The aim of this study is to confirm by a randomized double-blind controlled study the interest of a combination of saffron (Saffr'Activ®) and scutellaria (Scutell'up®) on the regulation of mood.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man, aged of 18 to 75 years;
* Participant presenting a depressive episode, according to the DSM-5 definition;
* Participant presenting a BDI ≥ 14 and ≤ 28 at the inclusion, corresponding to mild to moderate symptoms;
* Participant with a recent episode of depression (less than 2 years), not managed by antidepressant or psychotherapeutic treatment;
* Participant with a current depressive disorder not requiring, in the investigator's opinion, the initiation of antidepressant medication;
* Provision of signed and dated informed consent form;
* Stated willingness to comply with all study procedures and availability for the duration of the study;
* French speaker.

Exclusion Criteria:

* Participant with a depressive disorder of another nature or any other mental pathology (schizophrenia, bipolarity, addiction to alcohol or drugs...);
* Participant at risk of suicide (determined by the Investigator, or HAMD item 3 score > 2) or having made a suicide attempt in the last 5 years;
* Participant with depression for more than 2 years;
* Participant undergoing psychotropic treatment (current or in the month prior to inclusion) (neuroleptic, anxiolytic, hypnotic);
* Participant with a serious health problem for which the Investigator considers that it is not in the participant's interest to participate in the study;
* Participant using products containing piperine or millpertuis, or having a known effect on mood within the last 4 weeks;
* Pregnant or breastfeeding women, or those planning to become pregnant within the next 8 weeks;
* Participant with an allergy or contraindication to any component of the study drug;
* Participant unable to understand study information (mental or linguistic disability);
* Participant who is participating or has participated in the previous month in another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluated mood regulation | Baseline and 6 weeks
  observe a difference of the Beck Inventory Depression (BDI) score (adjusted for baseline), after 6 weeks of supplementation. All items are scored on a 4-point scale, ranging from 0 to 3.

SECONDARY OUTCOMES:
Evaluated mood regulation | 3 and 6 weeks of intervention and after 2 weeks after the end of intervention
  Beck Inventory Depression (BDI) score. All items are scored on a 4-point scale, ranging from 0 to 3.
Evaluated mood regulation | after 3 and 6 weeks of intervention and after 2 weeks after the end of intervention
  Hamilton depression rating scale (HAMD) score. HAMD is composed of 21 items. The scoring is based on the first 17 items. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Dormal, PhD, Study Chair — Université Catholique de Louvain; Louise Deldicque, Pr, Study Director — Université Catholique de Louvain; Laurent Simar, Dr, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université Catholique de Louvain, CICN, Ottignies-Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No